CLINICAL TRIAL: NCT06519669
Title: A Single-arm Clinical Study of Autologous Tumor-Infiltrating Lymphocyte (GT201 Injection ) for Treatment of Patients with Advanced Lung Cancer
Brief Title: Autologous Tumor-Infiltrating Lymphocyte Injection(GT201) for Treatment of Patients with Advanced Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-201-016
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Adult; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT201 treatment group (Experimental)
  Interventions: Biological: GT201 injection

INTERVENTIONS:
Biological: GT201 injection — GT201 injection to treat Advanced lung cancer

SUMMARY:
This study is a single arm, open design aimed at evaluating the safety and tolerability of Autologous Tumor-Infiltrating Lymphocyte (GT201 injection ) for treatment of patients with Advanced lung cancer,while evaluating pharmacokinetic characteristics and efficacy assessment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily join the study, signed informed consent form，willing and able to comply with the study protocol;
* 2. Age 18 to 70 years old;
* 3. Queue 1: Late stage non-small cell lung cancer without driver genes that have failed first-line systemic treatment;Queue 2: Small cell lung cancer with first-line systemic treatment failure;
* 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* 5. Expected survival time of ≥ 12 weeks;
* 6. Good function of vital organs;
* 7. Subjects entering this study due to disease progression must have an imaging record of disease progression before tumor sampling;
* 8. At least one measurable target lesion that meets the definition of RECIST v1.1 after tumor sampling.

Exclusion Criteria:

* 1.Patients with uncontrollable tumor-related pain as judged by the investigator; participants requiring analgesic medication must already have a stable analgesic regimen at the time of study entry; symptomatic lesions suitable for palliative radiotherapy should be completed prior to study entry;
* 2.Known mental illness, alcoholism, drug use or substance abuse;
* 3.Pregnant or lactating women; or women who are pregnant, breastfeeding, or planning to become pregnant within 1 year after cell infusion;
* 4.Those who have received other clinical trial drug treatment within 4 weeks before preconditioning by lymphodepletion,plan to participate in other clinical trial drug treatment during the study;
* 5.The investigators determine that other conditions that make the patient not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-07-18 (Estimated); Study Completion 2027-07-18 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 years
  To evaluate efficacy parameters such Objective Response Rate (ORR) per RECIST 1.1, as assessed by the Investigator
Incidence and severity of adcersed events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection（GT307) in patients with relapsed/metastatic advanced solid tumor as measured by the incidence and severity of adcersed events per CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No